CLINICAL TRIAL: NCT07314294
Title: A Randomized, Open-label, Phase II Study of EMB-01 in Patients With Recurrent/Metastatic Colorectal Cancer
Brief Title: Phase II Study of EMB-01 in Recurrent/Metastatic Colorectal Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai EpimAb Biotherapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMB01X204
Record Dates: First submitted 2025-12-04; First posted 2026-01-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMB-01 1600 mg once weekly (QW) (Experimental): EMB-01 1600 mg administered once weekly throughout the study
  Interventions: Drug: EMB-01 1600 mg administered once weekly throughout the study
- EMB-01 1600 mg once weekly (QW) for 6 weeks, then 1600 mg every 2 weeks (Q2W) (Experimental): EMB-01 1600 mg once weekly for the first 6 weeks, then 1600 mg every 2 weeks thereafter
  Interventions: Drug: EMB-01 1600 mg once weekly for 6 weeks, then every 2 weeks thereafter

INTERVENTIONS:
Drug: EMB-01 1600 mg administered once weekly throughout the study — Participants receive EMB-01 at a dose of 1600 mg administered once weekly (QW) throughout the study.
  Arms: EMB-01 1600 mg once weekly (QW)
Drug: EMB-01 1600 mg once weekly for 6 weeks, then every 2 weeks thereafter — Participants receive EMB-01 at a dose of 1600 mg administered once weekly (QW) for the first 6 weeks, followed by 1600 mg administered every 2 weeks (Q2W) thereafter.
  Arms: EMB-01 1600 mg once weekly (QW) for 6 weeks, then 1600 mg every 2 weeks (Q2W)

SUMMARY:
This study is testing different dosing schedules of EMB-01 in patients with advanced colorectal cancer whose disease has recurrent or progressed on previous treatments. Patients will be randomly assigned to one of two dosing schedules: EMB-01 once weekly, or once weekly for 6 weeks then every two weeks.

DETAILED DESCRIPTION:
This is a randomized, open-label Phase II dose-optimization study of EMB-01 in patients with metastatic colorectal cancer (CRC). The study will enroll patients with recurrent/metastatic KRAS/BRAF wild-type left-sided CRC who have progressed, relapsed, or become intolerant after first- or second-line systemic therapy. Patients will be stratified by prior anti-EGFR therapy and randomized 1:1 into two groups.

Group 1 will receive EMB-01 1600 mg once weekly (QW). Group 2 will receive EMB-01 1600 mg QW for the first 6 weeks, followed by 1600 mg once every two weeks (Q2W).

Tumor assessments will follow RECIST v1.1 using CT and/or MRI. Baseline imaging will be performed within 28 days before enrollment. During the study, imaging and efficacy assessments will occur every 6 weeks for the first 12 cycles, and every 3 cycles thereafter. All imaging procedures must be consistent with baseline. Assessments will be performed by the investigator, with retrospective independent review if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the informed consent form (ICF).
2. Male or female aged ≥ 18 years.
3. Histologically or cytologically confirmed unresectable or metastatic left-sided colorectal cancer (primary tumor from splenic flexure to rectum) with at least one measurable lesion according to RECIST v1.1.
4. ECOG performance status ≤ 1.
5. Willing to provide a fresh tumor biopsy sample or a stored sample obtained within the past 2 years.
6. Adequate organ function prior to the first study treatment.
7. Prior anti-cancer treatment:

   1. Must have progressed on or been intolerant to at least first- or second-line systemic therapy for metastatic colorectal cancer. Prior therapy must include fluoropyrimidine, oxaliplatin, and irinotecan-based chemotherapy, and bevacizumab with or without cetuximab. Patients should not have received TAS-102, fruquinitinib, or regorafenib.
   2. Any approved or investigational anti-cancer therapy (chemotherapy, immunotherapy, hormone therapy except for replacement therapy, testosterone, or oral contraceptives, biological therapy, targeted therapy) must be discontinued ≥ 4 weeks or 5 half-lives (whichever is shorter) before first study treatment.
   3. Palliative radiotherapy, bone metastasis radiotherapy, or oral fluoropyrimidines (e.g., tegafur, capecitabine) must be stopped ≥ 2 weeks before first study treatment; no therapeutic radiotherapy within 8 weeks before first EMB-01 dose.
8. Women of childbearing potential or male patients with partners of childbearing potential must use one or more contraceptive methods from clinical screening and continue during study treatment until 3 months after the last EMB-01 dose.

Exclusion Criteria:

1. Presence of KRAS/NRAS exon 2, 3, 4 mutations, BRAF V600 mutation, HER2 positivity (IHC3+ or amplification), dMMR/MSI-H, RET fusion, NTRK fusion, or other molecular mutations affecting anti-EGFR or cMET efficacy(Investigator and sponsor discussion recommended if applicable), based on central lab testing or prior treatment history.
2. Life expectancy < 3 months.
3. Residual adverse events (AEs) from prior anti-cancer therapy > CTCAE grade 1.
4. Primary CNS malignancy or symptomatic CNS metastases (brain, leptomeningeal, or arachnoid). Patients with asymptomatic CNS metastases may be eligible if no local radiotherapy is needed, or radiotherapy was completed ≥ 4 weeks prior to study treatment.
5. Pregnant or breastfeeding women.
6. Major surgery within 28 days prior to screening. Surgical wounds must be fully healed.
7. Idiopathic pulmonary fibrosis, unresolved active or chronic inflammatory lung disease, or history of interstitial lung disease (ILD). Patients with resolved radiation pneumonitis may be eligible.
8. History of Stevens-Johnson syndrome, toxic epidermal necrolysis, or severe skin infections.
9. Prior dual anti-EGFR and cMET therapy.
10. Prior EGFR inhibitor therapy discontinued due to severe skin toxicity.
11. Other significant medical conditions, psychiatric or psychological disorders, or familial/endemically high-risk diseases that may interfere with study assessments, treatment, follow-up, adherence, or increase risk of treatment-related complications.
12. Any condition deemed by the investigator to make study participation not in the patient's best interest or likely to interfere, limit, or confound study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Drom the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Objective response rate of EMB-01 at different dose levels
Number of participants with Adverse Events and Serious Adverse Events as assessed by CTCAE v5.0 | Screening up to follow-up (30 days after the last dose)
  Number of participants with Adverse Events and Serious Adverse Events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Best Overall Response (BOR) as assessed by RECIST v1.1 | from the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Best Overall Response (BOR) as assessed by RECIST v1.1
Cmax | Up to 3 months after first study drug administration
  PK parameter Cmax of EMB-01 at different dose levels
ADA | Up to the 30-day safety follow-up visit after EOT
  Incidence of anti-drug antibodies (ADA) of EMB-01 at different dose levels
Ctrough | Through treatment completion, an average of 1 year
  Measured trough concentration (Ctrough) of EMB-01
Area under the concentration-time curve from time 0 (pre-dose) to the time of the dosing interval (AUC0-t) | up to 3 months after first study drug administration
  Area under the concentration-time curve from time 0 (pre-dose) to the time of the dosing interval (AUC0-t)
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | up to 3 months after first study drug administration
  Area under the concentration-time curve from time 0 to infinity (AUC0-inf)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou

IPD SHARING:
Plan to Share IPD: No